CLINICAL TRIAL: NCT00350220
Title: A Prospective, Randomized, Controlled Clinical Trial Comparing Two Transfusion Strategies in Pediatric Patients Undergoing Cavopulmonary Connection.
Brief Title: Transfusion Strategies in Pediatric Cardiothoracic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, jill cholette, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12408
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2010-02-25 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-05

CONDITIONS: Congenital Heart Disease
Keywords: Single ventricle; Bidirectional Glenn; Fontan; Congenital cardiac disease; Red blood cell transfusion; oxygen utilization; lactate level; hemoglobin level
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart | interventions — Bloodless Medical and Surgical Procedures

ARMS (2):
- 1 (Active Comparator): High Hemoglobin group; goal Hb >13g/dl. 10cc/kg RBCs are transfused for any hemoglobin value under 13g/dl regardless whether clinical indication for transfusion exists.
  Interventions: Other: transfusion strategy
- 2 (Active Comparator): Low Hb transfusion group; goal to not transfuse unless the Hb <9.0 g/dl. 10cc/kg RBCs are transfused only if the Hemoglobin is under 9.0g/dl and clinical indications for transfusion exist.
  Interventions: Other: Low Hb transfusion group

INTERVENTIONS:
Other: transfusion strategy — For the High Hb group; transfusions will be given to keep the Hb >13.0 g/dl
  Arms: 1
Other: Low Hb transfusion group — RBCs will not be transfused unless the Hb < 9.0 g/dl
  Arms: 2

SUMMARY:
The purpose of this study is to determine the best red blood cell(hemoglobin) level for infants and children following surgical repair of particular heart defects. These children often receive red blood cell transfusions after surgery, but what the best hemoglobin level is for them remains unknown.

DETAILED DESCRIPTION:
Objective: To compare mean post-operative arterial lactate levels, oxygen utilization, and outcome measures in pediatric patients undergoing cavopulmonary connection managed with two different red blood cell transfusion strategies.

Methods: We propose a prospective, randomized clinical trial of sixty-six pediatric patients with cyanotic, complex congenital cardiac disease undergoing cavopulmonary connection as their operative repair. Thirty-three patients will be randomly assigned to a low Hb strategy of transfusion, in which red cells are transfused if the hemoglobin concentration falls below 9.0 g/dL, and hemoglobin concentrations are maintained about 8.5 g/dL. Thirty-three additional patients will be randomly assigned to the high Hb transfusion strategy, where red cells are transfused if the hemoglobin concentration falls below 13.0 g/dL, and hemoglobin concentrations are maintained about 12.5 g/dL. The primary endpoint will be comparison of mean arterial lactate levels from 8 to 72 hours post-operatively. The secondary endpoints will be oxygen utilization reflected by the arterio-venous oxygen difference (AV-difference) and arterio-cerebral oxygen difference (AC-difference). Measures of oxygen utilization will be derived from arterial oxygen saturation (SaO2), mixed venous oxygen saturation (SvO2), and cerebral oxygen saturation (ScO2) collected at various time points throughout the study. Tertiary outcome measures will be length of mechanical ventilation, length of oxygen use and of vasoactive agent administration, length pediatric cardiac intensive care unit (PCICU) admission, volume of blood transfused, and mortality. Data from each group will be compared using analysis of variance to assess for the presence of a difference between the two transfusion strategies. If a significant difference between the two groups exists, T-tests will be performed to compare data points between each group to assess for a significant difference.

Hypothesis: A more restrictive (low Hb) strategy of red cell transfusion will be as effective as, and possibly superior to, the historical (high Hb) approach. Allowing a lower Hb concentration will decrease RBC donor exposure and may decrease the known complications of RBC transfusions. We postulate that no significant difference will exist between the two transfusion groups in regards to hemodynamic and cardiopulmonary status (as evidenced by mean lactate levels) and oxygen utilization.

ELIGIBILITY:
Inclusion Criteria:

* 4 months to 6.99 years of age
* surgical candidates for cavopulmonary connection
* English speaking

Exclusion Criteria:

* presence of known bleeding disorder
* presence of known coagulopathy
* age < 4 months
* age > 7 years
* non-English speaking

Ages: 4 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Cholette, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449

RESULTS

PARTICIPANT FLOW:
Groups:
- High Hemoglobin (Liberal) Group: High Hemoglobin group; goal Hb >13g/dl. RBCs transfused for any Hemoglobin under 13g/dl regardless clinical indications for transfusion.
- Low Hb (Restrictive) Group: Low Hb transfusion group; RBCs are not transfused unless the Hb <9.0 g/dl and clinical indications for transfusion are met.
Period: Overall Study
Arm/Group | High Hemoglobin (Liberal) Group | Low Hb (Restrictive) Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Hemoglobin (Liberal) Group | Low Hb (Restrictive) Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants] — subjects under 8 years of age included
  Participants
    <=18 years | 30 | 30 | 60
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.75 (1.9) | 2.25 (1.8) | 2.5 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Lactate Level
Description: Mean arterial lactate for the first 48 hours post-op.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High Hemoglobin (Liberal) Group | Low Hb (Restrictive) Group
Number analyzed (Participants) | 30 | 30
mmol/L | 1.4 (0.4) | 1.4 (0.5)

2. Secondary Outcome: Oxygen Utilization During the 8 Hour to 72 Hours Post-operative Period.
Time Frame: 3 days
Reporting Status: Not Posted

3. Secondary Outcome: Length of Mechanical Ventilation
Time Frame: 3 days
Reporting Status: Not Posted

4. Secondary Outcome: Length of Oxygen Use
Time Frame: 3 days
Reporting Status: Not Posted

5. Secondary Outcome: Length of Vasoactive Agent Administration
Time Frame: 3 days
Reporting Status: Not Posted

6. Secondary Outcome: Volume of Blood Transfused
Time Frame: 3 days
Reporting Status: Not Posted

7. Secondary Outcome: Mortality Before Hospital Discharge
Time Frame: 30 days
Reporting Status: Not Posted

8. Primary Outcome: Peak Arterial Lactate Level
Description: Peak arterial lactate level for the 48 hour post-op study period.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | High Hemoglobin (Liberal) Group | Low Hb (Restrictive) Group
Number analyzed (Participants) | 30 | 30
mmol/l | 3.2 (1.3) | 3.1 (1.5)

ADVERSE EVENTS:
Arm/Group | High Hemoglobin (Liberal) Group | Low Hb (Restrictive) Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
There were no limitations to this study. There was 100% compliance with study procedures. There were no adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No